CLINICAL TRIAL: NCT02794337
Title: Integrated Phase II/III Randomized Control Trial of Transarterial Chemoembolisation Alone or in Combination With Stereotactic Body Radiation in Patients With Unresectable Hepatocellular Cancer
Brief Title: TACE vs TACE+SBRT for Unresectable Hepatocellular Cancer
Acronym: TACE-SBRT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Associate Professor, Radiation Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC IEC III 91
Record Dates: First submitted 2016-03-08; First posted 2016-06-09 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB TACE Arm (Active Comparator): Patients randomized to drug eluting beads(DEB) TACE arm will undergo 3 cycles of DEB-TACE (100 mg of doxorubicin drug eluting beads which will be repeated after 4-6 weeks. CT/MRI will be repeated prior to each cycle. Sorafenib will be omitted on the day of TACE and will be reinitiated after the TACE procedure. After completing all TACE cycles patients will continue to be on sorafenib till progression, or 12 months whichever is later, or in patients who fail to tolerate it after dose modifications. Hepatobiliary CTCAE will be completed at baseline, at each TACE cycle and subsequently at each follow up. QOL will be evaluated at the same time and also at two months after completing all sessions of TACE (matched time point with completion of SBRT in interventional arm)
  Interventions: Procedure: TACE; Drug: Sorafenib
- DEB-TACE+SBRT arm (Experimental): Patients randomized to DEB TACE/SBRT arm will undergo DEB-TACE as in standard arm. SBRT will be initiated 4-6 weeks after last TACE procedure. During this period patients will stop Sorafenib. SBRT once initiated will continue for 2-2.5 weeks. Sorafenib will be reinitiated 4 weeks after SBRT completion and will continue to be administered till progression or 12 months whichever is earlier, or in patients who fail to tolerate it after dose modifications. QOL will be evaluated at baseline, before each cycle of TACE, 1 month after SBRT and three monthly thereafter. Hepatobiliary CTCAE will be completed at baseline, after each TACE, before SBRT and after completion of SBRT and subsequently at each follow up.
  Interventions: Radiation: SBRT; Procedure: TACE; Drug: Sorafenib

INTERVENTIONS:
Radiation: SBRT — Intervention involves administering high precision radiation to the tumour in 6-8 fractions over 2-2.5 weeks
  Other Names: Stereotactic Ablative Radiation
  Arms: DEB-TACE+SBRT arm
Procedure: TACE — Involves catheterization of the tumour feeding vessels and injecting 100 mg of doxorubicin drug eluting beads. Maximum 3 TACE procedures are done
  Other Names: Transarterial chemoembolisation
Drug: Sorafenib — Sorafenib will be initiated 2 weeks before 1st TACE at a dose considered appropriate by the treating clinician. Though 400 mg bid is the recommended dose a lower dose may be used as per the judgement of treating clinician. It will be omitted on the days of TACE and SBRT. Sorafenib will be reinitiated 4 weeks after SBRT completion and will continue to be administered till progression or 12 months whichever is earlier. Sorafenib can however be stopped in patients who fail to tolerate sorafenib even after dose modifications.
  Other Names: Tyrosine Kinase Inhibitor

SUMMARY:
Vast majority of patients with hepatocellular carcinoma (HCC) present with unresectable disease. In the last decade results of randomized trials and a subsequent metaanalyses established transarterial chemoembolization (TACE) or systemic chemotherapy (sorafenib) as standard of care. However, TACE alone is not a curative approach. The two year survival following TACE ranges from 31-63% with almost 100% patients developing disease progression after treatment. There is need to investigate additional therapeutic options that would consolidate the initial response to TACE. A recent metaanalyses concluded that addition of high dose radiation to TACE results in 10-35% improvement in two year overall survival. However as results of metaanalyses were based on studies with small sample size, unclear randomization procedure and heterogenous dose of radiation, the need for conducting a high quality randomized study was highlighted The present study is designed to investigate the role of high dose conformal radiation as consolidation therapy after TACE in patients with nonmetastatic unresectable HCC.

DETAILED DESCRIPTION:
Resection or liver transplant is the only curative treatment in patients with hepatocellular carcinoma (HCC) however a vast majority of patients present with unresectable disease. In the last decade results of randomized trials and a subsequent metaanalyses established transarterial chemoembolization (TACE) as standard of care in patients with Barcelona Clinic Liver Cancer (BCLC) stage B. However, TACE alone is not a curative approach. The two year survival following TACE ranges from 31-63% with almost 100% patients developing disease progression after treatment. There is need to investigate additional therapeutic options that would consolidate the initial response to TACE. A recent metaanalyses including 17 trials (5 randomized and 12 non randomized studies) concluded that addition of high dose radiation to TACE results in upto 10-35% improvement in two year overall survival. However as results of metaanalyses were based on studies with small sample size, unclear randomization procedure and heterogenous dose of radiation, the need for conducting a high quality randomized study was highlighted. The present study is designed to investigate the role of high dose conformal radiation as consolidation therapy after TACE in patients with nonmetastatic unresectable HCC.

With an integrated phase II/III design the study investigates the impact of local radiation therapy on infield progression free survival in patients with locally advanced unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC. Tissue diagnosis is not mandatory however desirable. In the absence of tissue diagnosis imaging findings characteristic of HCC will be used. i.e. in high risk population a nodule with arterial phase enhancement and wash out during portovenous phase will be considered as diagnostic of HCC. In patients where one imaging is not conclusive another imaging modality will be used. However if second imaging is also inconclusive and Alpha Feto Protein (AFP) is within the nondiagnostic or borderline range than tissue diagnosis will be deemed mandatory.
* Barcelona Stage B/ Barcelona A not deemed suitable for Sx or refuse surgery. Child Pugh A/Select Child Pugh B (score7/10).
* Eastern Cooperative Oncology Group Performance Status 0-1.
* Total number of measurable target lesions 2 or less than 2, can be encompassed within a single hepatic field or 2 different hepatic fields without exceeding safe dose limit constraints.
* Optimal predicted liver volume reserve >700 cc. No Contraindication for TACE. Tumor considered to be sufficiently away from GI structures to deliver safe radiation dose (>1 cm).
* Willing for molecular banking of tumour tissue (optional).

Exclusion Criteria:

* Metastatic or nodal disease on staging investigations.
* Child C Cirrhosis or previous history of liver failure. Expected life span <6 months.
* Active variceal bleeding or other signs of hepatic decompensation.
* Portal venous thrombosis rendering patients unsuitable for TACE. However if pt is suitable for superselective TACE then can be considered for trial inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
In-field Progression Free Survival | Upto 24 months
  The trial is designed to assess a benefit in in-field progression free survival. The principal investigator would assess the study results 24 months after last accrual.

SECONDARY OUTCOMES:
Cause Specific Survival | Upto 24 months
  Will compare the cause specific survival between both the arms
Response assessment after treatment | Upto 24 months
  Using modified Response Evaluation Criteria in Solid Tumors scoring, radiological response to treatment will be assessed between both the arms.
Quality of Life Assessment of patients over a period of time | Upto 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) Study Group on Quality of Life has developed the Quality of life questionaires (QLQ) which are EORTC QLQ-C30 and the hepatocellular carcinoma specific EORTC QLQ-HCC 18 consisting in a modular system for assessing the quality of life of cancer patients in clinical research. EORTC QLQ-HCC 18 is an 18-item questionnaire designed to be used along with the 30-item EORTC QLQ-C30 Each item will be scored according to the EORTC guidelines
Toxicity Assessment | Upto 24 months
  Assessment will be done according to CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Chopra, MD, Principal Investigator — ACTREC,Tata Memorial Centre
Locations (2):
- India (2):
  - Advanced Centre for Treatment, Research and Education in Cancer, Tata Memorial Centre, Navi Mumbai, Maharashtra
  - Advanced Centre of Treatment Research and Education In Cancer,Tata Memorial Centre, Navi Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided